CLINICAL TRIAL: NCT03567603
Title: A Comparison of Mismatch Negativity Waveform Differences in Opioid-exposed and Non-exposed Neonates.
Brief Title: Sound Processing Changes in Babies With Opioid Exposure
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ronnie Guillet, Professor of Pediatrics, University of Rochester
Other Study IDs: RSRB#72329
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid exposed neonates: prenatal opioid exposure
- non-opioid exposed neonates: no prenatal opioid exposure

SUMMARY:
The purpose of this study is to identify problems with interpreting sounds in babies that have been exposed to opioids prior to birth. Being able to identify these issues in infancy may allow us to find children who may have problems with language learning later in life so that we can try to minimize these.

DETAILED DESCRIPTION:
This is a single center prospective study of neonates >36 weeks' gestation prenatally exposed to psychoactive substances and gestationally age-matched controls. Evoked response potentials on EEG in response to auditory oddball paradigms will be compared between cohorts. Analyses will try to identify differences in auditory processing using ANOVAs to compare the mismatch negativity measures, amplitudes and latencies as a function of study group.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 36 weeks, confirmation of dates via ultrasound or last menstrual period
* Prenatal opioid exposure ("exposed"), confirmed via admitted use or newborn drug screen; no prenatal opioid exposure ("control") by maternal report or testing
* All races, ethnicities, sexes to be included
* Informed permission form signed by mother

Exclusion Criteria:

* Birth weight ≤ 3rd percentile or ≥ 97th percentile for gestational age
* Have comorbid medical disorders including; those associated with sensorineural hearing loss, significant congenital anomalies, congenital heart disease, known brain injury/malformations
* Infants requiring mechanical ventilation
* Infants requiring continuous sedation

Max Age: 20 Days | Sex: All
Age Groups: Child
Study Population: Investigators with routine access to infant and maternal records will identify subjects based on review of patient charts upon admission to the NICU or nursery.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Percent with neonates with auditory cortical processing deficiencies | baseline
  A bone conducting sound playback lead will be placed over a bony prominence on the skull to transmit the auditory oddball paradigm that will be repeatedly played via this lead. The oddball paradigm will consist of a repeating sound loop including multiple identical 5-30 decibels tones of same duration interspersed with single 5-30 decibels tone of different pitch but same duration (deviant tone). Continuous EEG recordings will be collected during playback.
  EEG tracings will be analyzed specifically for the mismatch negativity waveforms. Comparisons will be made between the deviant and standard responses (sound tones) and the percentage of neonates with no difference between the standard and deviant waveforms will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Guillet, MD, PHD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No